CLINICAL TRIAL: NCT05396703
Title: Feasibility and Complications After Transoral Endoscopic Thyroidectomy Via Vestibular Approach (TOETVA) - a Single-Center First Experience Case Series and Systematic Review
Brief Title: TOETVA Feasibility and Complications - Single Center First Experience
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: BWO Z2021024
Record Dates: First submitted 2022-05-11; First posted 2022-05-31 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2022-05

CONDITIONS: Thyroid Gland Disease; Surgery
Keywords: TOETVA; NOTES; Surgery; Endocrine; Thyroid; Case Series
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TOETVA: All patients who underwent a transoral endoscopic thyroidectomy via vestibular approach (TOETVA) at the investigators' center.
  Interventions: Procedure: TOETVA

INTERVENTIONS:
Procedure: TOETVA — Completed procedure.

SUMMARY:
All participants who underwent (or will undergo) a transoral endoscopic thyroidectomy via vestibular approach (TOETVA) at the investigators' center are observed for complications and feasibility of this surgery. Anonymised data relevant to the participants' condition will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent (or will undergo) a transoral endoscopic thyroidectomy via vestibular approach (TOETVA) at the investigators' center

Exclusion Criteria:

* Patients who did not undergo (or will not undergo) a TOETVA at the investigators' center

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent (or will undergo) a transoral endoscopic thyroidectomy via vestibular approach at the investigators' center.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Complications initial | Immediately postoperative (during hospitalization)
  Complications after performed surgery
Complications before follow-up | If premature presentation occurs (admission after discharge and before follow-up consultation at 1 month after surgery)
  Complications after performed surgery
Complications before follow-up | Data at first follow-up visit will be reported. First follow-up visit will be at (average) 1 month after discharge.
  Complications after performed surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kinet, MD, Principal Investigator — Zuyderland MC
Locations (1):
- Zuyderland MC, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised patient sex, age, extent of resection, preoperative TSH values, TI-RADS classification, Bethesda classification, malignancy of lesion, and complications after surgery will be provided within the final manuscript.

REFERENCES:
- [Derived] Kinet S, van Weezelenburg MAS, Pijnenburg A, Stoot JHMB, van Bastelaar J. Feasibility and complications after transoral endoscopic thyroidectomy via vestibular approach (TOETVA) - a single-center first experience case series. Langenbecks Arch Surg. 2024 May 15;409(1):158. doi: 10.1007/s00423-024-03347-3. PMID 38748236